CLINICAL TRIAL: NCT03649074
Title: Software Treatment for Actively Reducing Severity of ADHD as Adjunctive Treatment to Stimulant (STARS-ADHD Adjunctive)
Brief Title: Software Treatment for Actively Reducing Severity of ADHD as Adjunctive Treatment to Stimulant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akili Interactive Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001S-A
Record Dates: First submitted 2018-08-23; First posted 2018-08-28 (Actual); Results first posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: The study will enroll participants into one of two cohorts according to stimulant status. Both cohorts will be assigned to AKL-T01 (with AKL-X01 symptom tracking).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- AKL-T01 (Experimental): AKL-T01 digital treatment.
  Interventions: Device: AKL-T01

INTERVENTIONS:
Device: AKL-T01 — AKL-T01 multitasking digital treatment. AKL-T01 multitasking treatment employs perceptual discrimination attention/memory task as well as a continuous motor "driving" task.

SUMMARY:
The purpose of this study is to determine the effects of combining AKL-T01 (with AKL-X01 symptom tracking) as adjunctive treatment to stimulant medication, and to understand the effects of AKL-T01 treatment (with AKL-X01 symptom tracking) in participants not recently on medication.

DETAILED DESCRIPTION:
The study aims to enroll (203) participants, with a confirmed diagnoses of ADHD, at approximately 15 sites and will be divided between 2 cohorts; 130 participants will be enrolled in Cohort 1, and 73 participants will be enrolled in Cohort 2.

Cohort 1 will have been stable (adherence to a prescribed medication schedule) on a stimulant medication, but are inadequately managed by the stimulant (in the opinion of the investigator). The stimulant is managed by their own physician for at least 30 days before baseline. This is the Stimulant cohort.

Cohort 2 will have been stable without any stimulant medication for at least 30 days before the baseline. This is the Non-Stimulant cohort.

For both cohorts, at least 7 and up to 30 days before baseline, participants' caretakers will begin using AKL-X01 (Fengo) to track their participants' symptoms and behaviors.

During Treatment Phase 1 (Days 1 through 28) participants in Cohort 1 (Stimulant) will continue to receive their current stimulant plus the addition of AKL-T01. Participants in Cohort 2 (Non-Stimulant) will just receive AKL-T01. For both cohorts, during this time the caretakers will monitor their child's symptoms daily with AKL-X01.

During the 1-Month Break (Days 29 through 56) between AKL-T01 treatment phases, participants in Cohort 1 will continue to receive their current stimulant. In both cohorts, AKL-T01 will be suspended during this time. For both cohorts, during this time caretakers will continue to monitor their child's symptoms daily with AKL-X01.

During Treatment Phase 2 (Days 57 through 84), participants in Cohort 1 (stimulant) will continue to receive their current stimulant plus the addition of AKL-T01. Participants in Cohort 2 will just receive AKL-T01. For both cohorts, during this time the caretakers will monitor their child's symptoms daily with AKL-X01.

AKL-T01, or EVO Multi, is a digital intervention that requires the subject to navigate a character through a game-like space, while collecting objects, in a fixed period of time.

AKL-T01: Videogame-like digital therapy

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ages 8 years 0 months to 14 years 9 months (inclusive), at the time of parental informed consent.
2. Confirmed ADHD diagnosis (primarily inattentive or combined subtype), at Screening based on DSM-V criteria and established via the MINI-KID administered by a trained clinician.

   Note: Co-morbid diagnoses on the MINI-KID are acceptable provided that ADHD is the primary diagnosis and the co-morbid diagnoses will not confound study data (per the Investigator's judgment).
3. Currently experiencing sub-optimal treatment of ADHD, based upon results of Clinical Global Impression-Severity score.
4. Impairment Rating Scale (Parent Report) score of ≥ 3 at Screening.
5. Ability to follow written and verbal instructions (English), as assessed by the PI and/or study coordinator.
6. Estimated IQ score > 80 as assessed by the Kaufmann Brief Intelligence Test, Second Edition (KBIT-II).
7. Ability to comply with all testing, requirements, study procedures, and availability for the duration of the study.
8. Provision of signed and dated parental informed consent form and assent form.
9. Participant's parent and/or caregiver has access any of the following Apple™ or Android™ smart phone and/or mobile devices (for accessing AKL-X01 application): Apple iPhone 6, 6+, 7, 8, 10; Android Samsung Galaxy S7, S7 Edge, S8, S8+, S9, S9+; Android Samsung Note 8; Android LG G6, G7, V30, K20. Apple mobile devices must be running iOS 11.2+. Android mobile devices must be running Nougat or Marshmallow.
10. For Cohort 1 (stimulant), participant must be stable** on stimulant medication, at an approved FDA dose , for ≥ 30 days prior to enrollment (may also be one stimulant plus a booster, provided that the dose is stable and does not change throughout the course of the trial).

    **Note: Medication stability is defined as:
    * Moderate response on stimulant, but still room for improvement
    * Dose unchanged within past 30 days, but other doses have been tried previously without improvement
    * Currently taking stimulant, but parent and/or caregiver wishes not to increase dosage for any reason
    * Taking consistent stimulant dose on weekdays, but not on weekends
11. For Cohort 2 (non-stimulant), participant must be stable off stimulant medication for ≥ 30 days prior to enrollment.

Exclusion Criteria:

1. Current, controlled (requiring a restricted medication) or uncontrolled, comorbid psychiatric diagnosis , based on MINI-KID and subsequent clinical interviewing, with significant symptoms including but not limited to:

   1. post-traumatic stress disorder
   2. psychosis
   3. bipolar illness
   4. pervasive developmental disorder
   5. severe obsessive compulsive disorder
   6. severe depressive
   7. severe anxiety disorder
   8. conduct disorder
   9. other symptomatic manifestations that in the opinion of the Investigator may confound study data/assessments.

   Participants with clinical history of learning disorders will be allowed to participate, provided the disorder does not impact their ability to participate in the trial based on PI judgment.
2. Participants who are currently treated with a non-stimulant medication for ADHD (i.e., atomoxetine, clonidine, guanfacine).
3. Participants diagnosed with ADHD Hyperactive-Impulsive subtype, based upon score on the MINI-KID interview.
4. Participants showing no room for improvement, or those refractory to non-intensive ADHD treatment.
5. Initiation within the last 4 weeks from the time of consent of behavioral therapy. Participants who have been in behavior therapy consistently for more than 4 weeks may participate provided their therapy frequency and intensity is unchanged during the course of the study. Participants planning on changing or initiating behavior therapy during the course of the study will be excluded.
6. Participant is currently considered a suicide risk in the opinion of the Investigator, has previously made a suicide attempt, or has a prior history of, or is currently demonstrating active suicidal ideation or self-injurious behavior as measured by C-SSRS at Screening.
7. Motor condition (e.g., physical deformity of the hands/arms; prostheses) that prevents playing the digital treatment as reported by the parent or observed by the investigator.
8. Recent history (within the past 6 months) of suspected substance abuse or dependence
9. History of seizures (exclusive of febrile seizures), or significant motor or vocal tics, including but not limited to Tourette's Disorder)
10. Has participated in a clinical trial within 90 days prior to Screening.
11. Diagnosis of or parent-reported color blindness (Confirmed in-clinic via ICBT)
12. Uncorrected visual acuity (confirmed in-clinic, via ability of participant to play the game, at Screening)
13. Regular use of psychoactive drugs (non-stimulant) that in the opinion of the Investigator may confound study data/assessments.
14. Any other medical, behavioral, or developmental condition that in the opinion of the investigator may confound study data/assessments.
15. Has a sibling also enrolled/currently participating in the same study. Siblings may participate in the study sequentially, but not at the same time.
16. Has previously been randomized in a study of Akili's videogame-like digital treatment.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 206 (Actual)
Dates: Start 2018-12-28 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lazkowitz, MD, PhD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Melmed Center, Scottsdale, Arizona
  - Center for Psychiatry and Behavioral Medicine, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Flannery JE, Hinshaw SP, Kollins SH, Stamatis CA. Secondary analyses of sex differences in attention improvements across three clinical trials of a digital therapeutic in children, adolescents, and adults with ADHD. BMC Public Health. 2024 Apr 29;24(1):1195. doi: 10.1186/s12889-024-18597-5. PMID 38685016

RESULTS

PARTICIPANT FLOW:
Groups:
- AKL-T01 - Stimulant Cohort: Stable (adherence to a prescribed medication schedule) on a stimulant medication, but are inadequately managed by the stimulant (in the opinion of the investigator). The stimulant is managed by their own physician for at least 30 days before baseline.
- AKL-T01 - No-Stimulant Cohort: Stable without any stimulant medication for at least 30 days before the baseline.
Period: Overall Study
Arm/Group | AKL-T01 - Stimulant Cohort | AKL-T01 - No-Stimulant Cohort
Started | 130 | 76
Completed (Completed study through Day 28) | 124 | 71
Not Completed | 6 | 5
Not completed — Lost to Follow-up | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Withdrawn by Parent/Guardian | 1 | 2
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled in both the Stimulant (n=130) and No Stimulant (n=76) cohorts.
Groups:
- Total: Total of all reporting groups
Arm/Group | AKL-T01 - Stimulant Cohort | AKL-T01 - No-Stimulant Cohort | Total
Number analyzed (Participants) | 130 | 76 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.6 (1.75) | 10.5 (1.82) | 10.6 (1.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 20 | 52
  Male | 98 | 56 | 154
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — More than one race/ethnicity may be selected for participants, if applicable. Total number of participants distributed across categories may be greater than the Number of Participants Analyzed.
  Participants
    White | 106 | 57 | 163
    Black or African American | 21 | 16 | 37
    American Indian or Alaska Native | 3 | 1 | 4
    Asian | 8 | 2 | 10
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Other | 0 | 4 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 130 | 76 | 206

OUTCOME MEASURES:

1. Primary Outcome: Impairment Rating Scale, Overall Impairment (Change From Baseline to Posttreatment) in Cohort 1: Stimulant
Description: The Impairment Rating Scale (IRS) is a parent-rated scale that assesses individualized areas of impairment for a child participant and asks parents to make a rating of how significantly these problems impact functioning across a range of domains (social, family, school, self-esteem). Parents describe the primary areas of difficulty for each child and then provide a rating (via a Visual Analog Scale) of how much the difficulties affect the different areas of functioning ranging from (1) "no problem; definitely does not need treatment or special services" to (7) "extreme problem; definitely needs treatment or special services." The total IRS is 8 items, the 8th rating overall impairment. A negative change indicated a decrease in overall impairment.
Time Frame: Day 0 to Day 28
Population: Participants in the ITT (all participants who received a device) for whom both Day 0 and Day 28 data was able to be collected in full. For the IRS, this population included all participants for whom the eighth item of the questionnaire was completed. In the Stimulant cohort, two participants had the eighth item incomplete.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- AKL-T01 - Stimulant Cohort: AKL-T01, or EVO Multi, is a digital intervention that requires the subject to navigate a character through a game-like space, while collecting objects, in a fixed period of time.
  The Stimulant Cohort included participants who were stable on a stimulant medication prior to enrollment and throughout the study.
Arm/Group | AKL-T01 - Stimulant Cohort
Number analyzed (Participants) | 128
score on a scale | -0.7 (1.04)

2. Primary Outcome: Impairment Rating Scale, Overall Impairment (Change From Baseline to Posttreatment) in Cohort 2: Non-Stimulant
Description: as for outcome 1
Time Frame: Day 0 to Day 28
Population: Participants in the ITT (all participants who received a device) for whom both Day 0 and Day 28 data was able to be collected in full. For the IRS, this population included all participants for whom the eighth item of the questionnaire was completed. In the No-Stimulant cohort, two participants had the eighth item incomplete.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- AKL-T01 - No-Stimulant Cohort: AKL-T01, or EVO Multi, is a digital intervention that requires the subject to navigate a character through a game-like space, while collecting objects, in a fixed period of time.
  The No-Stimulant Cohort included participants who were not taking a stimulant medication prior to enrollment and remained off of a stimulant medication throughout the study.
Arm/Group | AKL-T01 - No-Stimulant Cohort
Number analyzed (Participants) | 74
score on a scale | -0.5 (0.89)

3. Secondary Outcome: ADHD-RS Total (Change From Baseline to Posttreatment) - Cohort 1: Stimulant
Description: The ADHD-RS-IV is an 18-item, clinician-administered questionnaire for which a parent respondent rates the frequency of occurrence of ADHD symptoms and behaviors as defined by criteria outlined for ADHD in the DSM-IV. Each item is scored on a 4-point scale ranging from 0 (rarely or never) to 3 (very often) with total scores ranging from 0-54. A higher score indicates more severe ADHD symptoms and behaviors. A negative change in total score indicates improvement from Day 0 to Day 28.
Time Frame: Day 0 to Day 28
Population: Participants in the ITT (all participants who received a device) Stimulant Cohort from whom both Day 0 and Day 28 data was collected in full. For the ADHD-RS, this includes all participants for whom all 18 items were completed. In the Stimulant cohort, two participants were missing a response for at least one item of the ADHD-RS.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AKL-T01 - Stimulant Cohort
Number analyzed (Participants) | 128
score on a scale | -6.1 (7.18)

4. Secondary Outcome: ADHD-RS Total (Change From Baseline to Posttreatment) - Cohort 2: Non-Stimulant
Description: as for outcome 3
Time Frame: Day 0 to Day 28
Population: Participants in the ITT (all participants who received a device) No-Stimulant Cohort from whom both Day 0 and Day 28 data was collected in full. For the ADHD-RS, this includes all participants for whom all 18 items were completed. In the No-Stimulant cohort, two participants were missing a response for at least one item of the ADHD-RS.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AKL-T01 - No-Stimulant Cohort
Number analyzed (Participants) | 74
score on a scale | -7.4 (9.92)

5. Secondary Outcome: CGI-I (at Posttreatment) - Cohort 1: Stimulant
Description: The Clinical Global Impression Scale - Improvement (CGI-I) is a clinician's comparison of the participant's overall clinical condition at follow up to the overall clinical condition at baseline. The CGI-S is a 7-point scale where 1 = Very much improved, 2=Much improved, 3=Minimally improved, 4=No change, 5=Minimally worse, 6=Much worse, and 7=Very much worse.
  A score of 1, 2, or 3 would indicate overall improvement of ADHD severity.
Time Frame: Day 28
Population: Participants in the ITT (all participants who received a device) Stimulant Cohort from whom Day 28 data was collected in full. For the CGI-I, this includes all participants for whom the assessment was completed. In the Stimulant cohort, two participants were not assessed at Day 28.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AKL-T01 - Stimulant Cohort
Number analyzed (Participants) | 128
score on a scale | 3.3 (0.84)

6. Secondary Outcome: CGI-I (at Posttreatment) - Cohort 2: Non-Stimulant
Description: as for outcome 5
Time Frame: Day 28
Population: Participants in the ITT (all participants who received a device) No-Stimulant Cohort from whom Day 28 data was collected in full. For the CGI-I, this includes all participants for whom the assessment was completed. In the No-Stimulant cohort, two participants were not assessed at Day 28.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AKL-T01 - No-Stimulant Cohort
Number analyzed (Participants) | 74
score on a scale | 3.4 (0.83)

7. Secondary Outcome: Change TOVA Attention Composite Score (ACS) - Cohort 1: Stimulant
Description: TOVA ACS is a comparison of the subject's scores based on selected measures that persons with an independent diagnosis of ADHD frequently demonstrated. ACS is calculated from variability, response time (RT), and d' Prime using the following formula: ACS = RT Z score (Half 1) + D' Z score (Half 2) + variability Z score (Total) + 1.80 where RT is the average time it takes to respond correctly to a target, D' score is a response discriminability score reflecting the ratio of "hits" to "false alarms", and variability is a measure of consistency of speed of responding based on the standard deviation of the mean correct response times. ACS tells how similar the score is to the ADHD profile. A score of less than -1.8 indicates that the subject had similar performance to a normative ADHD population. A lower score indicates a more severe ADHD profile. The calculation for difference in TOVA ACS is ACS at Baseline (Day 0) minus ACS at Day 28.
Time Frame: Day 0 to Day 28
Population: Participants in the ITT (all participants who received a device) Stimulant Cohort from whom Day 0 and Day 28 data was collected in full. For the TOVA, this includes all participants for whom the TOVA was completed. In the Stimulant cohort, two participants did not have complete TOVA assessments at Day 0 or Day 28.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | AKL-T01 - Stimulant Cohort
Number analyzed (Participants) | 128
z-score | 0.2 (3.34)

8. Secondary Outcome: Change TOVA Attention Composite Score (ACS) - Cohort 2: Non-Stimulant
Description: as for outcome 7
Time Frame: Day 0 to Day 28
Population: Participants in the ITT (all participants who received a device) No-Stimulant Cohort from whom Day 0 and Day 28 data was collected in full. For the TOVA, this includes all participants for whom the TOVA was completed. In the No-Stimulant cohort, three participants did not have complete TOVA assessments at Day 0 or Day 28.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | AKL-T01 - No-Stimulant Cohort
Number analyzed (Participants) | 73
z-score | -0.5 (2.78)

ADVERSE EVENTS:
Time Frame: 84 Days
Arm/Group | AKL-T01 - Stimulant Cohort | AKL-T01 - No-Stimulant Cohort
All-Cause Mortality (participants affected / at risk) | 0/130 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/130 | 0/76
Other Adverse Events (participants affected / at risk) | 22/130 | 15/76
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AKL-T01 - Stimulant Cohort (N=130) | AKL-T01 - No-Stimulant Cohort (N=76)
Frustration tolerance decreased (Psychiatric disorders) | 15 | 12
Irritability (Psychiatric disorders) | 2 | 1
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 1
Dizziness (Nervous system disorders) | 1 | 1
Asthenopia (Eye disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Feeling Abnormal (General disorders) | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/74/NCT03649074/Prot_SAP_000.pdf